CLINICAL TRIAL: NCT00581438
Title: Actual Approach to Treatment of Haemophilia A and B in Spain
Brief Title: Study Evaluating Approach to Treatment of Haemophilia A and B in Spain
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 3082A-102378
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Approach Haemophilia A and B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Analyze the clinical and therapeutic approach to treatment of haemophilia A and B in habitual clinical practice conditions in Spain.

DETAILED DESCRIPTION:
Analyze the clinical and therapeutic approach to treatment of haemophilia A and B in habitual clinical practice conditions in Spain during the first 3 years since diagnosis.

Assess haemophilia A or B patient profile, study different kinds of hanitual clinical treatment of haemophilia A and B patients, and estimate the kind of treatment and dosage units used per year in patients under habitual clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A or B patients of any age
* Written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People known to have Haemophilia A or B
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Analyze the clinical and therapeutic approach to treament of haemophilia A and B in habitual clinical practice conditions in Spain during the first 3 years since diagnosis. | 3 months

SECONDARY OUTCOMES:
Assess haemophilia A or B patient profile, study different kinds of habitual clinical treatment of haemophilia A and B patients, and estimate the dosage units used per year in patients under habitual clinical practice conditions. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer